CLINICAL TRIAL: NCT01873027
Title: OPtical Frequency Domain Imaging vs. INtravascular Ultrasound in Percutaneous Coronary InterventiON (OPINION)
Brief Title: OPtical Frequency Domain Imaging vs. INtravascular Ultrasound in Percutaneous Coronary InterventiON
Acronym: OPINION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Wakayama Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRICVD1225; UMIN000010580 (Registry Identifier: UMIN Clinical Trials Registry)
Record Dates: First submitted 2013-05-26; First posted 2013-06-07 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Percutaneous Coronary Intervention; Optical Frequency Domain Imaging; Intravascular Ultrasound
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OFDI-guided PCI (Experimental): * OFDI-guided PCI and assessment by OFDI at pre-PCI and post-PCI
  * Follow-up contact at the time of hospital discharge, 8 months and 12 months after PCI.
  Interventions: Device: OFDI
- IVUS-guided PCI (Active Comparator): * IVUS-guided PCI and assessment by IVUS at pre-PCI and post-PCI
  * Follow-up contact at the time of hospital discharge, 8 months and 12 months after PCI.
  Interventions: Device: IVUS

INTERVENTIONS:
Device: OFDI — * OFDI-guided PCI and assessment by OFDI at pre-PCI and post-PCI
  * Follow-up contact at the time of hospital discharge, 8 months and 12months after PCI
  Other Names: LUNAWAVE; Fastview; Biolimus a9-eluting stent (Nobori stent)
  Arms: OFDI-guided PCI
Device: IVUS — * IVUS-guided PCI and assessment by IVUS at pre-PCI and post-PCI
  * Follow-up contact at the time of hospital discharge, 8 months and 12months after PCI
  Other Names: VISIWAVE; ViewIT; Biolimus A9-eluting stent (Nobori stent)
  Arms: IVUS-guided PCI

SUMMARY:
The aim of this randomized study is to evaluate the impact of Optical frequency domain imaging (OFDI) guidance for Percutaneous Coronay Intervention (PCI) with drug-eluting stent (DES) as compared with Intravascular ultrasound (IVUS) guidance.

DETAILED DESCRIPTION:
Optical frequency domain imaging (OFDI) is a novel, high resolution intravascular imaging modality. Intravascular ultrasound (IVUS) is a widely used conventional imaging modality for achieving optimal stent deployment.

The aim of this randomized study is to evaluate the impact of OFDI guidance for Percutaneous Coronay Intervention (PCI) with drug-eluting stent (DES) as compared with IVUS guidance.

We will enroll 800 patients with a de novo lesion who will undergo PCI with DES as is routine practice. Patients will be rondomely assigned to either OFDI-guided PCI arm or IVUS-guided PCI arm.

Patients will then have a follow-up contact at the time of hospital discharge, 8 month and 12 month after PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a de novo lesion (in the native coronary circulation) and planned to undergo drug-eluting stent implantation for indications according to the Japan and USA guidelines
* Patients aged between 20 and 85 years old
* Patients who has provided written informed consent

Exclusion Criteria:

* Patients with Acute Myocardial Infarction (AMI) within 3 months
* Patients with cardiogenic shock
* Patients with chronic heart failure
* Patients with renal failure (eGFR <= 30 ml/min/1.73 m2 or Serum creatinine level >=1.5mg/dL)
* Patients who are currently enrolled in other clinical trial which has possibility to influence the primary endpoint of OPINION trial.
* Patients planned use of bare metal stent
* Patients with 3-vessel diseases
* Planned surgery within 1 year
* Patient on dialysis
* Target lesion such as:

  * Left main coronary artery
  * Aorto-Ostial lesion location within 3mm of the aorta junction
  * Chronic total occlusion
  * Small vessel (reference vessel diameter <2.5mm)
  * Coronary artery bypass graft

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 829 (Actual)
Dates: Start 2013-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Target Vessel Failure (TVF) | 12 months after PCI
  The composite endpoint comprised of cardiac death, target vessel-related myocardial infarction (MI) and clinically-driven target vessel revascularization (TVR)

SECONDARY OUTCOMES:
Cardiac death | 12 months after PCI
Myocardial Infarction (MI) | 12 months after PCI
Clinically-driven Target lesion revascularization (TLR) | 12 months after PCI
MACE (composite of cardiac death, MI, TLR) | 12 months after PCI
Target Vessel Revascularization (TVR) | 12 months after PCI
Stroke | 12 months after PCI
Stent thrombosis | 12 months after PCI
Binary restenosis | 12 months after PCI
Renal dysfunction | 8 months after PCI

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Akasaka, MD, PhD, Principal Investigator — Wakayama Medical University
Locations (1):
- Wakayama Medical University, Wakayama, Wakayama, Japan

REFERENCES:
- [Derived] Kubo T, Shinke T, Okamura T, Hibi K, Nakazawa G, Morino Y, Shite J, Fusazaki T, Otake H, Kozuma K, Ioji T, Kaneda H, Serikawa T, Kataoka T, Okada H, Akasaka T; OPINION Investigators. Optical frequency domain imaging vs. intravascular ultrasound in percutaneous coronary intervention (OPINION trial): one-year angiographic and clinical results. Eur Heart J. 2017 Nov 7;38(42):3139-3147. doi: 10.1093/eurheartj/ehx351. PMID 29121226